CLINICAL TRIAL: NCT00441103
Title: A Two-arm, Randomized, Double-blind, Control Group-compared, Multicenter, Phase IIIb Study With Monthly MRI and Biomarker Assessments to Evaluate the Efficacy, Safety, and Tolerability of Rebif® New Formulation (IFN Beta-1a) in Subjects With Relapsing Remitting Multiple Sclerosis
Brief Title: A Study to Evaluate Rebif® New Formulation (Interferon-beta-1a) in Relapsing Remitting Multiple Sclerosis
Acronym: IMPROVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 27178; 2006-003037-32
Record Dates: First submitted 2007-02-26; First posted 2007-02-28 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-06

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Subjects with relapsing remitting multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — peginterferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Rebif® New Formulation (IFN-beta-1a, RNF) (Experimental)
  Interventions: Drug: Rebif® New Formulation (IFN-beta-1a, RNF)
- Placebo/RNF (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Rebif® New Formulation (IFN-beta-1a, RNF)

INTERVENTIONS:
Drug: Rebif® New Formulation (IFN-beta-1a, RNF) — RNF will be administered at a dose of 44 mcg subcutaneously three times a week for 40 weeks.
  Other Names: IFN-beta-1a
  Arms: Rebif® New Formulation (IFN-beta-1a, RNF)
Drug: Placebo — Matching placebo will be administered subcutaneously three times a week for 16 weeks.
  Arms: Placebo/RNF
Drug: Rebif® New Formulation (IFN-beta-1a, RNF) — RNF will be administered at a dose of 44 mcg subcutaneously three times a week from Week 17 to Week 40.
  Other Names: IFN-beta-1a
  Arms: Placebo/RNF

SUMMARY:
General Note: throughout this record, "Rebif® New Formulation" is used for historical and consistency purposes.

Objectives:

Primary: To evaluate the efficacy of Rebif® New Formulation (Interferon-beta-1a [IFN-beta-1a], RNF), compared to placebo, in subjects with Relapsing Remitting Multiple Sclerosis and active disease by means of Magnetic Resonance Imaging (MRI) at the end of 16 weeks of treatment Secondary: To evaluate the efficacy of RNF by comparing the mean number of combined unique (CU) lesions per scan per subject between the initial 16 weeks of placebo treatment and 24 weeks of RNF treatment in the same subjects, originally randomized to placebo.

Primary Endpoints: The primary endpoint is the difference between the number of CU active MRI lesions at Week 16 in the RNF group (Group 1) versus the placebo group (Group 2).

Secondary Endpoints: The secondary endpoint is the difference in the mean number of CU active MRI lesions per scan per subject over the following treatment periods: Study Day 1 - Week 16 versus Weeks 17 - 40 for the subjects randomized to Group 2.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 60 years of age
* Female subjects must be neither pregnant nor breast-feeding and must lack child-bearing potential, as defined by either: post-menopausal or surgically sterile or use an effective method of contraception for the duration of the study
* Have Relapsing Remitting Multiple Sclerosis (RRMS) according to the revised McDonald criteria 2005
* Have brain and/or spinal MRI with findings typical of Multiple Sclerosis (MS)
* Have disease duration for more than 12 months
* Have disease activity characterized by at least one clinical event and one or more Gadolinium-enhancing MRI lesions within the 6 months prior to randomization
* Have score of <=5.5 on the Expanded Disability Status Scale (EDSS)
* Be willing and able to comply with the protocol for the duration of the study
* Have given written informed consent prior to any study-related procedure not part of the normal medical practice

Exclusion Criteria:

* Have any disease other than MS that could better explain his/her signs and symptoms
* Have complete transverse myelitis or bilateral optic neuritis
* Have received or have used anytime monoclonal antibodies, mitoxantrone, cytotoxic or immunosuppressive therapy (excluding systemic steroids and adrenocorticotrophic hormone [ACTH]), or total lymphoid irradiation
* Have received within 3 months prior to baseline any approved disease-modifying therapy for MS, cytokine or anti-cytokine therapy, intravenous immunoglobulin, plasmapheresis, any investigational drug, or experimental procedure
* Have received within 30 days prior to baseline oral or systemic corticosteroids or ACTH
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2006-12; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Stubinski, MD, Study Director — Merck Serono SA - Geneva, an affiliate of Merck KGaA Darmstadt, Germany

REFERENCES:
- [Result] De Stefano N, Curtin F, Stubinski B, Blevins G, Drulovic J, Issard D, Shotekov P, Gasperini C; IMPROVE Study Investigators. Rapid benefits of a new formulation of subcutaneous interferon beta-1a in relapsing-remitting multiple sclerosis. Mult Scler. 2010 Jul;16(7):888-92. doi: 10.1177/1352458510362442. Epub 2010 Mar 3. PMID 20200197
- [Result] De Stefano N, Sormani MP, Stubinski B, Blevins G, Drulovic JS, Issard D, Shotekov P, Gasperini C. Efficacy and safety of subcutaneous interferon beta-1a in relapsing-remitting multiple sclerosis: further outcomes from the IMPROVE study. J Neurol Sci. 2012 Jan 15;312(1-2):97-101. doi: 10.1016/j.jns.2011.08.013. Epub 2011 Aug 31. PMID 21880336
- [Derived] Giorgio A, Battaglini M, Gentile G, Stromillo ML, Gasperini C, Visconti A, Paolillo A, De Stefano N. Mapping the Progressive Treatment-Related Reduction of Active MRI Lesions in Multiple Sclerosis. Front Neurol. 2020 Nov 20;11:585296. doi: 10.3389/fneur.2020.585296. eCollection 2020. PMID 33329329
- See also: Full FDA approved prescribing information can be found here — http://www.mslifelines.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first participant first visit: 15 Dec 2006. Date of last participant last visit: 28 Nov 2008. Twenty five trial centers enrolled participants in the following countries: Bulgaria (7), Canada(2), Estonia (2), Germany (1), Italy(2), Lithuania (1), Romania (1), Russian Federation (4), Serbia (2), and Spain (3).
Pre-assignment Details: Participants meeting the eligibility criteria during screening period of up to 14 days were randomly assigned in a 2:1 ratio to receive either Rebif® New Formulation or matching placebo for 16 weeks. There were 33 screening failures: participants who did not meet all eligibility criteria (n=29), withdrawal of consent (n=3), and lost of view (n=1).
Groups:
- Rebif® New Formulation (IFN-beta-1a, RNF): RNF 44 microgram (mcg) administered subcutaneously three times a week for 40 weeks.
- Placebo/RNF: Matching placebo administered subcutaneously three times a week for 16 weeks, followed by RNF 44 mcg administered subcutaneously three times a week for subsequent 24 weeks.
Period: Overall Study
Arm/Group | Rebif® New Formulation (IFN-beta-1a, RNF) | Placebo/RNF
Started | 120 (Intent to treat (ITT) population: all participants who received at least one dose of study drug.) | 60 (Intent to treat (ITT) population: all participants who received at least one dose of study drug.)
Completed | 109 | 56
Not Completed | 11 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Death | 1 | 0
Not completed — Disease Progression | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Participant unable to use Rebiject II | 1 | 0
Not completed — Participant refused MRI | 1 | 0
Not completed — Inclusion criteria absent | 1 | 0
Not completed — Non-compliant | 0 | 1
Not completed — Participant decided to withdraw | 1 | 0
Not completed — Participant's reason | 0 | 1
Not completed — Participant decided to stop | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all randomized participants who received at least one dose of study drug.
Groups:
- Rebif® New Formulation (IFN-beta-1a, RNF): RNF 44 mcg administered subcutaneously three times a week for 40 weeks.
- Total: Total of all reporting groups
Arm/Group | Rebif® New Formulation (IFN-beta-1a, RNF) | Placebo/RNF | Total
Number analyzed (Participants) | 120 | 60 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 120 | 60 | 180
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (7.8) | 35.2 (10.5) | 34.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 42 | 130
  Male | 32 | 18 | 50
Region of Enrollment [Number; unit: participants]
  Bulgaria | 40 | 12 | 52
  Canada | 3 | 3 | 6
  Estonia | 8 | 5 | 13
  Germany | 1 | 0 | 1
  Italy | 7 | 4 | 11
  Lithuania | 5 | 3 | 8
  Romania | 11 | 8 | 19
  Russian Federation | 20 | 12 | 32
  Serbia | 20 | 9 | 29
  Spain | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Combined Unique (CU) Active Magnetic Resonance Imaging (MRI) Lesions at Week 16
Description: CU active lesions were defined as a unique newly active or persistently active lesion on the protocol density/time constant 2 (PD/T2) scan or the gadolinium (Gd-) enhanced time constant 1 (T1) scan (with a method to avoid double counting).
Time Frame: 16 Weeks
Population: ITT population included all randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Rebif® New Formulation (IFN-beta-1a, RNF) | Placebo/RNF
Number analyzed (Participants) | 120 | 60
lesions | 0.9 (1.4) | 3.0 (4.1)
Statistical Analysis 1: Comparison: Rebif® New Formulation (IFN-beta-1a, RNF) vs Placebo/RNF; Test type: Superiority or Other; p < 0.001, ANOVA — Non-parametric analysis of variance (ANOVA) with effects for treatment and the absence/presence of Gd-enhancing lesions at baseline as factors

2. Secondary Outcome: Mean Number of CU Lesions Per Scan Between the Initial 16 Weeks of Placebo Treatment and 24 Weeks of RNF Treatment in the Same Participants, Originally Randomized to Placebo.
Description: CU active lesions were defined as a unique newly active or persistently active lesion on the PD/T2 scan or the gadolinium enhanced T1 scan (with a method to avoid double counting). Only "Placebo Followed by RNF" arm was evaluable for this outcome measure.
Time Frame: Day 1 up to Week 16 and Week 17 up to Week 40
Population: ITT population included all randomized participants who received at least one dose of study drug. Here, "N" (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo/RNF
Number analyzed (Participants) | 57
lesions
  Day 1 up to Week 16 | 2.31 (2.63)
  Week 17 up to Week 40 | 0.65 (0.95)
Statistical Analysis 1: Comparison: Placebo/RNF; Mean difference was calculated by subtracting 'Day 1 up to Week 16' from 'Week 17 up to Week 40' and analyzed using Wilcoxon signed-rank test; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test; Mean Difference (Final Values) = -1.67, Standard Deviation 2.33

3. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. AEs were categorized based upon the treatment period during which they occurred, that is, double-blind period (up to Week 16) and rater-blind period (Week 17 up to Week 40).
Time Frame: Baseline up to Week 40
Population: Safety population included all randomized participants who received at least one dose of study drug. Here, 'n' signifies those participants who were evaluable for the specified category.
Measure: Number; unit: participants
Arm/Group | Rebif® New Formulation (IFN-beta-1a, RNF) | Placebo/RNF
Number analyzed (Participants) | 120 | 60
participants
  AEs during double-blind period (n = 120, 60) | 100 | 39
  AEs during rater-blind period (n = 112, 57) | 72 | 43
  SAEs during overall period (n = 120, 60) | 4 | 3

4. Secondary Outcome: Number of CU Active MRI Lesions
Description: CU active lesions were defined as a unique newly active or persistently active lesion on the PD/T2 scan or the gadolinium enhanced T1 scan (with a method to avoid double counting).
Time Frame: Up to Week 40
Population: ITT population included all randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Rebif® New Formulation (IFN-beta-1a, RNF) | Placebo/RNF
Number analyzed (Participants) | 120 | 60
lesions | 0.62 (1.29) | 1.27 (1.33)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 40
Arm/Group | Rebif® New Formulation (IFN-beta-1a, RNF) | Placebo/RNF
Serious Adverse Events (participants affected / at risk) | 4/120 | 3/60
Other Adverse Events (participants affected / at risk) | 100/120 | 39/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rebif® New Formulation (IFN-beta-1a, RNF) (N=120) | Placebo/RNF (N=60)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rebif® New Formulation (IFN-beta-1a, RNF) (N=120) | Placebo/RNF (N=60)
Influenza like illness (General disorders) | 60 (110) | 10 (10)
Injection site erythema (General disorders) | 39 (60) | 4 (6)
Injection site pain (General disorders) | 12 (13) | 1 (1)
Pyrexia (General disorders) | 9 (14) | 3 (5)
Asthenia (General disorders) | 8 (11) | 3 (8)
Chills (General disorders) | 8 (11) | 1 (3)
Fatigue (General disorders) | 7 (8) | 0 (0)
Headache (Nervous system disorders) | 37 (66) | 10 (17)
Dizziness (Nervous system disorders) | 3 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 7 (7) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (7) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (4)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other